CLINICAL TRIAL: NCT06580171
Title: A Study to Assess The Balance Using Remote Access Method - Walking and Remembering Test Validation
Brief Title: Validation of Walking and Remembering Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Assistant Professor (Principal Investigator), Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 25.07.2024/112
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Healthy Individuals
Keywords: Healthy; Walking and Remembering Test; Validity; Tele-assessment
MeSH Terms: interventions — Walking

STUDY DESIGN:
Intervention Model Description: Walking and Remembering Test Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking and Remembering Group (Experimental): Only Walking and Remembering Test will be applied to the group.
  Interventions: Other: Walking and Remembering Test

INTERVENTIONS:
Other: Walking and Remembering Test — Only Walking and Remembering Test will be applied to the group.

SUMMARY:
In this study, the usability of the Walking and Remembering Test will be examined using the remote interview method. The study will be carried out with a single group. First, the WART test will be performed face-to-face at Marmara University Biomechanics Laboratory. The second evaluation will be carried out using a remote method. From the participants;

* He/she will first be asked to walk freely within a line that is 8 meters long and 19 cm wide. Later;
* He will be asked to walk once at average speed and three times as fast as possible in the same line. Later;
* The participant is given a Counting Test. This test includes number sequences from 4 digits to 9 digits. Participants are told these number strings and asked to repeat them with the same speed and tone of voice. The longest sequence of numbers is recorded. Later;
* The participant is walked on the same line again and asked to repeat the longest number sequence he remembers and the test is completed. Cognitive performance with the counting test reflects walking speed during 4 walks, and the number of incorrect steps reflects walking performance.

ELIGIBILITY:
Inclusion Criteria:

* Having any known psychological, vestibular and neurological diseases,
* No major or minor hip, knee or ankle injuries,
* Not showing osteoarticular or muscle traumas that prevent upright posture and ambulation,
* Not taking medications that affect posture, such as vestibular apparatus sedatives, antidepressants or anxiolytics,
* Not complaining of dizziness or vertigo,
* Being between the ages of 18-30.

Exclusion Criteria:

* Individuals with untreated visual impairment,
* Epilepsy, postural dizziness or hypotension,
* Individuals with dependent ambulation,
* Individuals with any disease that affects balance,
* Those with cancer or fibromyalgia.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Walking and Remembering Test (WART) | Baseline of the study (Face-to-Face)
  WART is a clinical measure of dual-task ability involving individual and simultaneous motor and cognitive task performance. In the test, walking and memory are observed independently and under dual-task conditions.
Walking and Remembering Test (WART) | First day after the Baseline Assessment (Remote Assessment)
  WART is a clinical measure of dual-task ability involving individual and simultaneous motor and cognitive task performance. In the test, walking and memory are observed independently and under dual-task conditions.

SECONDARY OUTCOMES:
Demographic Data Form | Baseline of the study
  This form was created by researchers and it consist of personal informations such as gender, dominant extremity, history of sport, age, body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yildiz Ozer, Professor, Study Chair — Marmara University; Semra Oğuz, Associate Professor, Study Chair — Marmara University; Gökçe Kartal, MSc, Study Chair — Marmara University
Locations (1):
- Marmara University, Department of Physiotherapy and Rehabilitation, Biomechanics and Performance Analysis Laboratory, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No